CLINICAL TRIAL: NCT03265132
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Efficacy and Safety Study of 2 Dose Levels of Subcutaneous Anakinra (Kineret®) in Patients With Still's Disease (SJIA and AOSD)
Brief Title: A Study to Evaluate Efficacy and Safety of Anakinra in the Treatment of Still's Disease (SJIA and AOSD)
Acronym: anaSTILLs
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Meeting enrolment target (81 pat) will not be feasible within reasonable time.
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sobi.ANAKIN-301
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Results first posted 2020-04-28 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Still's Disease, Adult-Onset; Still's Disease, Juvenile-Onset
Keywords: Interleukin 1 receptor antagonist; IL-1 receptor antagonist; Kineret; anakinra; Adult-Onset Still's Disease; Systemic Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Still's Disease, Adult-Onset; Arthritis, Juvenile | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- anakinra (Experimental): 2 mg/kg/day (max 100 mg/day) or 4 mg/kg/day (max 200 mg/day)
  Interventions: Biological: anakinra
- Placebo (Placebo Comparator): Corresponding volume to anakinra 2 mg/kg/day or 4 mg/kg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: anakinra — sub cutaneous injection
  Other Names: Kineret
  Arms: anakinra
Drug: Placebo — sub cutaneous injection
  Arms: Placebo

SUMMARY:
The aim of this study is to demonstrate the efficacy and to evaluate the safety, pharmacokinetics (PK) and immunogenicity of anakinra in patients with newly diagnosed Still's disease, including SJIA (Systemic juvenile idiopathic arthritis) and AOSD (Adult-onset Still's disease).

DETAILED DESCRIPTION:
The study consists of a 12-week, randomized, double-blind, placebo controlled period with two dose levels of anakinra and a 4-week safety follow-up after last dose of investigational medicinal product (IMP). The primary endpoint will be evaluated at Week 2. Sustained efficacy and time to study drug discontinuation will be evaluated during the full study period.

A screening visit is optional and may be done to identify patients that could be suitable for the study. During the study 6 visits and 2 telephone contacts are scheduled i.e., Day 1 (baseline visit), Day 4Tel, Week 1, Week 2, Week 4, Week 8, Week 12 and Week 16Tel (End of Study).

Patients will be randomly assigned to study drug, after they meet all of the inclusion criteria and none of the exclusion criteria. Patients will receive treatment for 12 weeks, either anakinra or placebo. Patients will be randomized to anakinra in a dose of either 2 or 4 mg/kg/day, with a maximum dose of 100 or 200 mg once daily, respectively. Patients will be randomized to placebo with corresponding volumes for each of the two anakinra dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male and female patients with a body weight ≥ 10 kg.
3. Diagnosis of Still's disease.
4. If currently on glucocorticoid treatment, a stable dose for at least 1 week prior to randomization.
5. If currently on methotrexate treatment, a stable dose for at least 8 weeks prior to randomization.
6. Active disease.
7. Female patients of childbearing potential must use an effective method of contraception during the study (abstinence being a possible option) as well as present a negative pregnancy test prior to randomization.
8. Negative interferon-gamma release assay or Purified protein derivative ( PPD) test within 2 months prior to randomization. If not available, a test should be performed at day of randomization.

Exclusion Criteria:

1. Diagnosis of Still's disease more than 6 months prior to randomization.
2. Previous randomization into this study.
3. Participation in another concurrent clinical interventional study within 30 days of randomization.
4. Treatment with an investigational drug within 5 half-lives prior to randomization.
5. Previous or current treatment with anakinra, canakinumab or any other IL-1 inhibitor.
6. Use of the following therapies prior to randomization:

   * Narcotic analgesics within 24 hours prior to randomization.
   * Dapsone or etanercept within 3 weeks prior to randomization.
   * Intraarticular, intramuscular or intravenous administration of glucocorticoids or intravenous immunoglobulin (Ig) within 4 weeks prior to randomization.
   * Intravenous Ig with proven Still's disease modifying effect, leflunomide, infliximab or adalimumab within 8 weeks prior to randomization.
   * Thalidomide, cyclosporine, mycophenolate mofetil, 6-mercaptopurine, azathioprine, cyclophosphamide, chlorambucil or any other immunosuppressant within 12 weeks prior to randomization.
   * Tocilizumab within 12 weeks prior to randomization or any other immunomodulatory medication within 4 half-lives prior to randomization
   * Rituximab within 26 weeks prior to randomization.
7. Live vaccines within 1 month prior to randomization.
8. Known presence or suspicion of active, chronic or recurrent bacterial, fungal or viral infections, including tuberculosis, HIV infection or hepatitis B or C infection.
9. Clinical evidence of liver disease or liver injury.
10. Presence of severe renal function impairment.
11. Presence of neutropenia.
12. Presence or suspicion of MAS at baseline.
13. A diagnosis of MAS within the last 2 months prior to randomization.
14. History of malignancy within 5 years.
15. Known hypersensitivity to E coli-derived proteins, or any components of Kineret® (anakinra).
16. Pregnant or lactating women.
17. Foreseeable inability to cooperate with given instructions or study procedures.
18. Presence of any medical or psychological condition or laboratory result that in the opinion of the investigator can interfere with the patient's ability to comply with the protocol requirements or makes the patient not appropriate for inclusion to the study and treatment with IMP.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Ohlman, MD PhD, Study Director — Swedish Orphan Biovitrum
Locations (39):
- United States (36):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Attune Health, Beverly Hills, California
  - Rady Children's Hospital & Health Center, San Diego, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Mercy Hospital and Clinics, Kansas City, Kansas
  - University of Louisville School of Medicine Research Foundation, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Saint Paul Rheumatology, Eagan, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Institute for Rheumatic and Autoimmune Diseases, Summit, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Wake Forest Baptist Brenner Medical Center, Winston-Salem, North Carolina
  - MetroHealth System, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Univ of TX Southwestern Medical Center Dallas - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - University of Calgary - Alberta Children's Hospital, Calgary
  - University of Calgary, Calgary
  - The Hospital for Sick Children, Toronto

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 6 | 6 (One patient failed disease specific inclusion criteria and was excluded from efficacy analysis)
Completed | 6 | 0
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Progressive disease | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Anakinra | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (13.2) | 12.3 (19.3) | 13.3 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
Still's disease symptom duration [Mean (Standard Deviation); unit: Days] | 32.4 (18.7) | 109.0 (78.0) | 74.2 (69.1)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of ACR30 Responders With Absence of Fever Attributable to the Disease During the 7 Days Preceding Week 2.
Description: ACR30 response is defined as an improvement of ≥ 30% from baseline in at least 3 of any 6 variables listed below. Also no more than 1 of the 6 variables may worsen by >30% from baseline. (ACR: American College of Rheumatology)
  1. Physician global assessment of disease activity - Assessed on a Visual Analogue Scale (VAS) from no disease activity (0 mm) to very severe disease activity (100 mm).
  2. Patient/parent global assessment of overall well-being - Assessed on a VAS from very well (0 mm) to very poor (100 mm).
  3. Number of joints with active arthritis.
  4. Number of joints with limitation of motion.
  5. Assessment of physical function - Patient Reported Outcome instruments : Childhood Health Assessment Questionnaire (CHAQ) /Stanford Health Assessment Questionnaire (SHAQ).
  6. C-Reactive Protein (CRP) (mg/L).
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0022, Fisher Exact; Risk Difference (RD) = 1.0, 95% CI 2-sided [0.42 to 1.00]

2. Secondary Outcome: Proportion of ACR30 Responders With Absence of Fever During 24 Hours Preceding Week 1.
Description: ACR30 response is defined as an improvement of ≥ 30% from baseline in at least 3 of any 6 variables listed in the description of the primary outcome measure. Also no more than 1 of the 6 variables may worsen by >30% from baseline.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 5 | 3

3. Secondary Outcome: Proportion of ACR50 Responders With Absence of Fever During 24 Hours Preceding Week 1.
Description: ACR50 response is defined as an improvement of ≥ 50% from baseline in at least 3 of any 6 variables listed in the description of the primary outcome measure. Also no more than 1 of the 6 variables may worsen by >30% from baseline.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 5 | 2

4. Secondary Outcome: Proportion of ACR70 Responders With Absence of Fever During 24 Hours Preceding Week 1.
Description: ACR70 response is defined as an improvement of ≥ 70% from baseline in at least 3 of any 6 variables listed in the description of the primary outcome measure. Also no more than 1 of the 6 variables may worsen by >30% from baseline.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 5 | 0

5. Secondary Outcome: Proportion of ACR90 Responders With Absence of Fever During 24 Hours Preceding Week 1.
Description: ACR90 response is defined as an improvement of ≥ 90% from baseline in at least 3 of any 6 variables listed in the description of the primary outcome measure. Also no more than 1 of the 6 variables may worsen by >30% from baseline.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 4 | 0

6. Secondary Outcome: Proportion of ACR50 Responders With Absence of Fever During 7 Days Preceding Week 2.
Description: as for outcome 3
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 0

7. Secondary Outcome: Proportion of ACR70 Responders With Absence of Fever During 7 Days Preceding Week 2.
Description: ACR70 response is defined as an improvement of ≥ 70% from baseline in at least 3 of any 6 variables listed in the description of the primary outcome. Also no more than 1 of the 6 variables may worsen by >30% from baseline.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 0

8. Secondary Outcome: Proportion of ACR90 Responders With Absence of Fever During 7 Days Preceding Week 2.
Description: ACR90 response is defined as an improvement of ≥ 90% from baseline in at least 3 of any 6 variables listed in the description of the primary outcome . Also no more than 1 of the 6 variables may worsen by >30% from baseline.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 5 | 0

9. Secondary Outcome: Proportion of Responders in Physician Global Assessment of Disease Activity.
Description: Assessed on a VAS from no disease activity (0 mm) to very severe disease activity (100 mm). Response is defined as an improvement of ≥ 30%, 50%, 70% and 90% from baseline. Only improvement of ≥90% at Week 2 reported here.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 4 | 0

10. Secondary Outcome: Proportion of Responders in Patient/Parent Global Assessment of Overall Well-being.
Description: Assessed on a VAS from very well (0 mm) to very poor. (100 mm). Response is defined as an improvement of ≥ 30%, 50%, 70% and 90% from baseline.Only improvement of ≥90% at Week 2 reported here.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 4
Participants | 4 | 0

11. Secondary Outcome: Proportion of Responders in Number of Joints With Active Arthritis.
Description: Response is defined as an improvement of ≥ 30%, 50%, 70% and 90% from baseline.Only improvement of ≥90% at Week 2 reported here.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 3 | 2

12. Secondary Outcome: Proportion of Responders in Number of Joints With Limitation of Motion.
Description: as for outcome 11
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 4 | 2

13. Secondary Outcome: Proportion of Responders in Assessment of Physical Function (CHAQ/SHAQ).
Description: Childhood Health Assessment Questionnaire (CHAQ) and Stanford Health Assessment Questionnaire (SHAQ) assess physical and functional status (see Clinical protocol section 6.5.4.1.5). Response is defined as an improvement of ≥ 30%, 50%, 70% and 90% from baseline. Only improvement of ≥90% at Week 2 reported here.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 4 | 0

14. Secondary Outcome: Proportion of Responders in CRP (mg/L).
Description: Response is defined as an improvement of ≥ 30%, 50%, 70% and 90% from baseline. Only improvement of ≥90% at Week 2 reported here.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 5 | 0

15. Secondary Outcome: Proportion of Patients With Absence of Fever During the 7 Days Preceding Week 2.
Description: Proportion of patients with absence of fever during the 7 days preceding Week 2.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 0

16. Secondary Outcome: Proportion of Patients With Absence of Fever During the 24 Hours Preceding Week 1.
Description: Absence of fever during the 24 hours preceding week 1.
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 4

17. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Week 1.
Description: Change from baseline in Physician global assessment of disease activity measured on a VAS 0 (very well)-100 (very poor) at Week 1.
Time Frame: Day 1 and Week 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
mm | -46.3 (32.6) | -30.0 (18.5)

18. Secondary Outcome: Change From Baseline in Patient/Parent Global Assessment of Overall Well-being at Week 1.
Description: Change from baseline in patient/parent global assessment of overall well-being measured on a VAS 0 (very well)-100 (very poor) at Week 1.
Time Frame: Day 1 and Week 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 4
mm | -53.7 (27.7) | -25.0 (31.7)

19. Secondary Outcome: Change From Baseline in CRP.
Description: Change from baseline in C-Reactive Protein (CRP). CRP is measured in mg/L.
Time Frame: Day 1 and Week 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
mg/L | -109.6 (63.4) | -22.7 (47.1)

20. Secondary Outcome: Proportion of Patients With Sustained ACR30, ACR50, ACR70 and ACR90 Response.
Description: Proportion of patients that still meet the corresponding week 2 response with absence of fever in the preceding 7 days. Only the strictest criteria, ACR90, is reported here.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 6 | 0

21. Secondary Outcome: Proportion of Patients With Sustained ACR30, ACR50, ACR70 and ACR90 Response in Relation to Glucocorticoid Tapering.
Description: Please note no patients were treated with any systemic glucocorticoids at randomization. Hence no results available.
Time Frame: Week 2, Week 4, Week 8 and Week 12
Population: No patients were treated with any systemic glucocorticoids at randomization
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Proportion of Patients With Absence of Rash.
Description: Absence of rash is evaluated 24 hours preceding Week 1 and 7 days preceding Week 2, Week 4, Week 8 and Week 12. Only data at Week 2 reported here.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 4
Participants | 5 | 2

23. Secondary Outcome: Change From Baseline in CRP.
Description: Change from baseline in CRP. Results at Week 2 reported here.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
mg/L | -126.670 (66.697) | -33.904 (64.393)

24. Secondary Outcome: Change From Baseline in Hemoglobin (Hb). Results at Week 2 Reported Here.
Description: Change from baseline in Hemoglobin (Hb). Results at Week 2 reported here.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 3
g/dL | 1.57 (0.86) | -0.80 (1.01)

25. Secondary Outcome: Change From Baseline in Platelet Count.
Description: Change from baseline in platelet count. Results at Week 2 reported here.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 3
10^9/L | -148.2 (52.3) | -26.3 (139.6)

26. Secondary Outcome: Change From Baseline in Ferritin.
Description: Change from baseline in ferritin. Results at Week 2 reported here.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 5 | 3
ug/L | -390.364 (387.521) | -49.383 (51.776)

27. Secondary Outcome: Change From Baseline in Patient/Parent Global Assessment of Disease Related Pain.
Description: Assessed on a VAS from no pain (0 mm) to very severe pain (100 mm).
Time Frame: Week 2
Population: Patients with baseline and week 2 data analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 4
score on a scale | -55.6 (27.7) | -33.5 (28.5)

28. Secondary Outcome: Time to Study Drug Discontinuation for Any Reason.
Description: Time to study drug discontinuation was analyzed using Kaplan-Meier curves. Number of patients with premature study drug discontinuation for any reason is reported here.
Time Frame: From Day 1 to Week12
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 0 | 5

29. Secondary Outcome: Time to Study Drug Discontinuation Due to Lack of Efficacy or Progressive Disease.
Description: Proportion of study drug discontinuation due to lack of efficacy or progressive disease was analyzed using Kaplan-Meier curves. Number of patients discontinuing study drug due to lack of efficacy or progressive disease is reported here.
Time Frame: From Day 1 to Week12
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 0 | 4

30. Secondary Outcome: Proportion of Patients Who Have Initiated Tapering of Glucocorticoids.
Description: Please note no patients were treated with any systemic glucocorticoids at randomization. Hence no results available
Time Frame: From Week 2 to Week12
Population: No patients were treated with any systemic glucocorticoids at randomization
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Proportion of Patients That Have Decreased the Glucocorticoid Dose With at Least 50% From Baseline.
Description: Please note no patients were treated with any systemic glucocorticoids at randomization. Hence no results available
Time Frame: From Week 2 to Week12
Population: No patients were treated with any systemic glucocorticoids at randomization
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Percentage Decrease of the Glucocorticoid Dose From Baseline.
Description: Please note no patients were treated with any systemic glucocorticoids at randomization. Hence no results available
Time Frame: From Day 1 to Week12
Population: No patients were treated with any systemic glucocorticoids at randomization
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Proportion of Patients With at Least One Adverse Event.
Description: All adverse events collected from start of study treatment up to 28 days after stopping study treatment.
Time Frame: From Day 1 to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 6 | 4

34. Secondary Outcome: Proportion of Patients With at Least One Serious Adverse Event Including Death.
Description: Serious adverse events (SAEs) will be collected from informed consent up to 28 days after stopping study treatment.
Time Frame: From Informed consent to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 0 | 1

35. Secondary Outcome: Proportion of Patients With Macrophage Activation Syndrome (MAS).
Description: Proportion of patients with Macrophage Activation Syndrome (MAS).
Time Frame: From Day 1 to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

36. Secondary Outcome: Proportion of Patients With Antidrug Antibodies (ADA) Against Anakinra.
Description: Proportion of patients with antidrug antibodies (ADA) against anakinra.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 6 | 1

37. Secondary Outcome: Proportion of Patients With Neutralizing Antibodies.
Description: Confirmed ADA positive samples will be analyzed for the presence of neutralizing antibodies.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

38. Secondary Outcome: Anakinra Serum Pre-dose Concentrations.
Description: Week 2 reported here.
Time Frame: Week 2
Population: No data available for the placebo group as they did not receive anakinra.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 4 | 0
ng/mL | 157 (134) |

39. Secondary Outcome: Anakinra Serum Pharmacokinetic Parameters: Cmax,
Description: PK parameters only available for 2 patients.
Time Frame: Week 12
Population: PK parameters only available for 2 anakinra treated patients.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Anakinra
Number analyzed (Participants) | 0 | 2
ng/mL |  | 1990.0 (1315.2)

40. Secondary Outcome: Anakinra Serum Pharmacokinetic Parameters, Tmax and T½
Description: PK parameters only available for 2 patients
Time Frame: Week 12
Population: PK parameters only available for 2 patients
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Anakinra
Number analyzed (Participants) | 0 | 2
hours
  Tmax |  | 3.06 (1.33)
  T½ |  | 5.23 (1.01)

41. Secondary Outcome: Anakinra Serum Pharmacokinetic Parameter: AUC 0-24 h
Description: PK parameters only available for 2 patients
Time Frame: Week 12
Population: PK parameters only available for 2 anakinra treated patients
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Placebo | Anakinra
Number analyzed (Participants) | 0 | 2
h*ng/mL |  | 18483.3 (15708.4)

42. Secondary Outcome: Anakinra Serum Pharmacokinetic Parameter: CL/F
Description: Pharmacokinetic parameters only available for 2 patients
Time Frame: Week 12
Population: Pharmacokinetic parameters only available for 2 anakinra treated patients
Measure: Mean (Standard Deviation); unit: mL/h*kg
Arm/Group | Placebo | Anakinra
Number analyzed (Participants) | 0 | 2
mL/h*kg |  | 170.80 (45.69)

43. Secondary Outcome: Anakinra Serum Pharmacokinetic Parameter: Vd/F
Description: PK parameters only available for 2 patients
Time Frame: Week 12
Population: PK parameters only available for 2 anakinra treated patients
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Placebo | Anakinra
Number analyzed (Participants) | 0 | 2
mL/kg |  | 1254.52 (95.57)

44. Secondary Outcome: Change From Baseline in JADAS27.
Description: Juvenile Arthritis Disease Activity Score (JADAS) includes 4 measures: physician global assessment of disease activity, patient or parent global assessment of overall well-being, 27 active joint count, and CRP. The JADAS27 includes the 27 joints. JADAS27 is calculated as the sum of its four components, physician global assessment of disease activity converted to cm from the VAS (0=no activity, 10=maximum activity); patient global assessment of well-being converted to cm from the VAS (0=very well, 10=very poor); active joint count (0-27); and CRP. Prior to calculation CRP is truncated to a 0 - 10 scale according to the following formula: (CRP (mg/l) -10)/10. Before calculation, CRP values <10 mg/l are converted to 10 and CRP values >110 mg/l are converted to 110. The JADAS27 tool yields a global score of 0-57.
  Only results from Week 2 reported here.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 4
score on a scale | -21.42 (3.93) | -15.81 (4.83)

45. Secondary Outcome: Number of Days Off School or Work Due to Still's Disease.
Description: Number of days off school or work due to Still's disease week 1-2.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 4
Days | 0.7 (1.6) | 1.3 (2.5)

46. Secondary Outcome: Proportion of Patients With Inactive Disease.
Description: Inactive disease is a composite of the following parameters: no joints with active arthritis, no fever, no rash, no serositis, no splenomegaly, no generalized lymphadenopathy attributable to Still's disease, CRP level within normal limits, physician's global assessment of disease activity score below 10 mm on a 100 mm VAS and a documented morning stiffness ≤15 minutes.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 3 | 0

47. Secondary Outcome: Change From Baseline in IL-6.
Description: Only results from Week 2 reported here.
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 3
ng/L | -30.048 (23.262) | -24.818 (25.940)

48. Secondary Outcome: Change From Baseline in IL-18.
Description: Only results from Week 2 reported here
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 5 | 3
ng/L | -7968.0 (7564.4) | -20701.7 (32766.4)

49. Secondary Outcome: Change From Baseline in Serum Calprotectin.
Description: Change from baseline in serum calprotectin. Only results from Week 2 reported here
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 6 | 3
mg/L | -100.038 (113.349) | -26.021 (23.819)

50. Secondary Outcome: Change From Baseline in Neopterin.
Description: Only results from Week 2 reported here
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 5 | 3
nmol/L | -3.08 (5.69) | -8.00 (10.82)

ADVERSE EVENTS:
Time Frame: From the start of study treatment up to 28 days after stopping study treatment.
Description: The Investigator recorded all directly observed AEs, and all AEs spontaneously reported by the patient, in the CRF. MAS was defined as an event of special interest in this study. If a MAS diagnosis was made at any point after patient signed informed consent, the event was to be reported as a serious AE and the patient should be withdrawn from the study.
Arm/Group | Anakinra | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=6) | Placebo (N=6)
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=6) | Placebo (N=6)
Upper respiratory infection (Infections and infestations) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Vitamin D decrease (Investigations) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03265132/Prot_001.pdf
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT03265132/SAP_000.pdf